CLINICAL TRIAL: NCT03237104
Title: Back in the Game: A Pilot Study Assessing an Immediate Functional Progression Program in Athletes With a Spondylolysis.
Brief Title: Back in the Game: An Immediate Functional Progression Program in Athletes With a Spondylolysis.
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Mitchell Selhorst, Physical Therapist/Principle Investigator, Nationwide Children's Hospital
Other Study IDs: IRB17-00258
Record Dates: First submitted 2017-07-31; First posted 2017-08-02 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Low Back Pain; Spondylosis
Keywords: Adolescent; Athlete
MeSH Terms: conditions — Low Back Pain; Spondylosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute spondylolysis: Athletes who meet the inclusion criteria and consent to participate in the pilot study will be referred directly to PT care for 2 times per week until cleared to return to sport.
  Interventions: Other: Immediate PT

INTERVENTIONS:
Other: Immediate PT — Athletes will perform phase I (neutral spine) of the program and progress to phase II (functional motion) as able without an increase in pain and without compensations noted in function. The athlete will be assessed at each session to determine if they meet the criteria to begin the next step of functional progression program. Once the athlete has met the criteria of phase II, they will progress into the final phase of the functional progression program for return to sport activity. As these athletes progress through the third phase, and are able to meet the return to sport criteria, they will be released to return to sport. Athletes will not be released to return to sport prior to their first physician follow-up visit at 4 weeks.

SUMMARY:
Half of all adolescents report experiencing low back pain (LBP), and adolescents who are active in sport report an even higher rate. The most common identifiable cause of LBP in the adolescent athlete is a stress fracture in the low back, known as a spondylolysis. Spondylolysis injuries have been found in up 47% of young athletes with LBP. The current recommendations of care for a spondylolysis consist of rest for at least 3 months, bracing, and physical therapy. These recommendations result in athletes being out of sport for as long as 46 months, and are based on low level evidence and expert opinion. In addition to the long period out of sport, 42% have poor long-term outcomes, and 1 in 6 athletes are no longer able to play at their former level specifically due to their back injury. These long periods out of sport and poor long-term clinical outcomes suggest current care recommendations are suboptimal.

The overall objective of the proposed research is to test the feasibility of using an early functional progression program to reduce athletes' time out of sport and improve clinical outcomes. Specifically, to pilot altering the rest period in athletes with a spondylolysis and begin rehabilitation immediately. These young athletes will return to sport as they are able, after demonstrating predetermined pain free functional ability. Twelve young athletes with a confirmed active spondylolysis will be recruited to undergo the early function progression intervention. The specific aims of this study are to assess the feasibility of implementing the immediate functional progression protocol, refine the protocol if necessary, and estimate potential effectiveness of this intervention. The athletes' outcomes will be compared to historical controls. The investigators hypothesize that the immediate functional progression program can be successfully implemented and with only minor changes will be suitable for use in larger trials. It is estimated the immediate functional progression program has the potential to return athletes to sport more than a month sooner than current practice. Once able to demonstrate the feasibility of the early functional progression program, the investigators plan to progress this work into larger trials to fully assess effectiveness, safety and long-term outcomes.

DETAILED DESCRIPTION:
Athletes who meet the inclusion criteria and consent to participate in the pilot study will be referred directly to physical therapy (PT) care for 2 times per week. Athletes will follow-up with their co-investigating physician every 4 weeks until discharge. The immediate functional progression program will be performed by physical therapists trained in the treatment protocol. Athletes will perform phase I of the program and progress to phase II as able without an increase in pain and without compensations noted in function. The athlete will be assessed at each session to determine if they meet the criteria to begin the next step of functional progression program. Once the athlete has met the criteria of phase II, they will progress into the final phase of the functional progression program for return to sport activity. As these athletes progress through the third phase, and are able to meet the return to sport criteria, they will be released to return to sport. Athletes will not be released to return to sport prior to their first physician follow-up visit at 4 weeks.

Phase I Immediate Functional Progression Program Core strengthening in neutral spine Treat directional preference if identified Hip strengthening Peri-scapular strengthening Flexibility exercises Manual Therapy as needed Modalities for pain (use sparingly)

Phase II Immediate Functional Progression Program Core strengthening in functional range Hip and peri-scapular strengthening Flexibility exercises Manual Therapy (use sparingly) Phase III Immediate Functional Progression Program- Return to Sport Return to sport activity with focus on functional return to all aspect of sport.

Signs of not responding as anticipated during the immediate functional progression program: Inability to meet long-term goals of care in PT including inability to return to sport due to low back pain within three months, an increase in pain or no significant decrease in pain (<2/10) at physician visits until patient reports <2/10 pain with activity.

Sample Size A sample size of 12 will be recruited for this pilot trial. As there is a nonlinear relationship between confidence interval (CI) width and sample size, further increases in participants beyond 12 have a diminishing benefit on precision for preliminary studies.

Data Analysis Descriptive statistics of the patient demographics and outcome variables will be reported. Inferential calculations will not be performed as this is a pilot to demonstrate the feasibility of implementing the proposed immediate functional progression program.

Aim 1: Discussion of the success of implementing the immediate functional progression program will occur during and after care of each patient. The PI will monitor patient documentation to assess adherence to the research protocol in care. Adverse events will be monitored, the immediate functional progression program will be considered acceptably tolerated by patients if <3 adverse events are observed.

Aim 2: (Potential Problems and Alternative strategies) Minor problems identified in the pilot study will serve to refine to the protocol for the full randomized clinical trial. Larger potential problems include non-adherence to the experimental treatment protocol. The risk of this potential problem will be reduced by training of all staff involved in the research process. If a problem is found in the experiment protocol that inhibits patients from satisfactorily progressing in their care, the co-investigators will meet and decide on a course of action to fix this issue. An alteration in the experimental protocol that results in improved care would be considered a positive outcome, as the goal of this pilot study is to demonstrate viability and feasibility for a larger clinical trial.

Aim 3: Clinical outcomes including pain, function, time to return to sport and recurrence of symptoms will be compared against historical controls to assess for potential efficacy. Historical controls for quality of life are not available in this population. Time to return to sport will be the primary outcome of interest. A decrease in return to sport time of > 30 days compared to the historical control time of 3.8 months without a notable worsening of other outcomes will indicate future research is warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Age 10-19 years old
2. Diagnosed with a spondylolysis through magnetic resonance imaging (MRI) with active signs of healing. Signs of active healing are defined as edema noted on MRI.
3. Participates in organized sport

Exclusion Criteria:

1. Previous rest from activity >4 weeks without improved symptoms
2. Red flags present (bowel/bladder problems, saddle anesthesia, progressive neurological deficits, recent fever or infection, unexplained weight loss, unable to change symptoms with mechanical testing)
3. Numbness and tingling in any lumbar dermatome
4. Other injury or condition that would alter the plan of care for spondylolysis (i.e. pregnancy, anterior cruciate ligament (ACL) tear, concussion)
5. History of lumbar surgery

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population of interest is young athletes with a recent spondylolysis injury.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Time to return to sport (days) | 1-6 months
  The number of days from diagnosis of spondylolysis to the point the patient passes all criteria of the PT program and is cleared to return to sport by the physician

SECONDARY OUTCOMES:
Change in Micheli Functional Scale (MFS) | Baseline, 1 month, 3 months, 6 months, 1 year
  Function
Change in Numeric Pain Rating Scale | Baseline, 1 month, 3 months, 6 months, 1 year
  Pain
Recurrence of low back symptoms | Baseline, 1 month, 3 months, 6 months, 1 year
  Patients will be asked if there low back pain (must have impaired ability to play sport or activities of daily living)
adverse reaction | 1-6 months
  An adverse reaction will be defined as 1) lumbar symptoms increasing enough to cause an unplanned visit to a physician or 2) the patient being placed on hold from therapy during the episode of care
Change in MRI | Baseline, 3 months
  Patients will have a repeat MRI performed at 3 months. A radiologist will assess for change in the spondylolytic lesion, edema and anterolisthesis.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Nationwide Children's Hospital Sports and Ortho PT Ortho Center, Columbus, Ohio
  - Nationwide Children's Hospital Sports and Ortho PT East Broad, Columbus, Ohio
  - Nationwide Children's Hospital Sports and Ortho PT Dublin, Dublin, Ohio
  - Nationwide Children's Hospital Sports and Ortho PT New Albany, New Albany, Ohio
  - Nationwide Children's Hospital Sports and Ortho PT Westerville, Westerville, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anderson K, Sarwark JF, Conway JJ, Logue ES, Schafer MF. Quantitative assessment with SPECT imaging of stress injuries of the pars interarticularis and response to bracing. J Pediatr Orthop. 2000 Jan-Feb;20(1):28-33. PMID 10641684
- [Background] Klein G, Mehlman CT, McCarty M. Nonoperative treatment of spondylolysis and grade I spondylolisthesis in children and young adults: a meta-analysis of observational studies. J Pediatr Orthop. 2009 Mar;29(2):146-56. doi: 10.1097/BPO.0b013e3181977fc5. PMID 19352240
- [Result] Selhorst M, Fischer A, Graft K, Ravindran R, Peters E, Rodenberg R, Welder E, MacDonald J. Timing of Physical Therapy Referral in Adolescent Athletes With Acute Spondylolysis: A Retrospective Chart Review. Clin J Sport Med. 2017 May;27(3):296-301. doi: 10.1097/JSM.0000000000000334. PMID 27347866
- [Result] Selhorst M, Fischer A, Graft K, Ravindran R, Peters E, Rodenberg R, MacDonald J. Long-Term Clinical Outcomes and Factors That Predict Poor Prognosis in Athletes After a Diagnosis of Acute Spondylolysis: A Retrospective Review With Telephone Follow-up. J Orthop Sports Phys Ther. 2016 Dec;46(12):1029-1036. doi: 10.2519/jospt.2016.7028. Epub 2016 Nov 8. PMID 27825292